CLINICAL TRIAL: NCT03870477
Title: Intracapsular and Intertrochanteric Fracture Fixation With the THP Hip Fracture Plating System
Brief Title: THP Hip Fracture Plating System Study
Acronym: THP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to remove product from portfolio.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSU2017-22T
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Femur Fracture; Femur Fracture Intertrochanteric; Garden Grade I Subcapital Fracture of Femoral Neck; Garden Grade II Subcapital Fracture of Femoral Neck; Garden Grade III Subcapital Fracture of Femoral Neck; Garden Grade IV Subcapital Fracture of Femoral Neck
Keywords: Cannulated Screws; Lag Screws; Compression Screws; Telescoping Lag Screws; Cortical Screws; Hip Fracture Plate
MeSH Terms: conditions — Femoral Fractures; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- THP Hip Fracture Plating System (Other): THP Hip Fracture Plating System in Intracapsular and Intertrochanteric Femur Fractures
  Interventions: Device: THP Hip Fracture Plating System with telescoping lag screws

INTERVENTIONS:
Device: THP Hip Fracture Plating System with telescoping lag screws — The fracture plates are contoured plates used in conjunction with telescoping lag screws that are 7.5mm in diameter with lengths ranging from 70mm to 130mm in 5mm increments.

SUMMARY:
The objective of this study is to systematically document the clinical outcomes of THP Hip Fracture Plating System when used to treat intracapsular and intertrochanteric fractures.

DETAILED DESCRIPTION:
Primary Endpoint:

• Revision rate due to device related complication(s) or non-union of the femur.

Secondary Endpoints:

• Radiographic and clinical fracture healing of the proximal femur using standard scoring methods.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient must be eligible for an open reduction and internal fixation of the proximal femur.
* Patient must have an intracapsular or intertrochanteric fracture.
* Patient must have need for alignment, stabilization, and reduction of bone fractures.
* Patient must have ability and willingness to follow postoperative care instructions until healing is complete.
* Patient must be in good nutritional state.
* Patient must be able and willing to sign the IRB/EC approved informed consent.

Exclusion Criteria:

* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Patient is known to be pregnant or breastfeeding.
* Patient has a psychiatric illness or cognitive deficit that will not allow proper informed consent.
* Infection.
* Patient conditions including bloody supply limitations, obesity or insufficient quantity or quality of bone.
* Patient with mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions.
* Patient has foreign body sensitivity. Where material sensitivity is suspected or unknown, testing is to be completed prior to implantation of the device.
* Patient is expected to be non-compliant with recommended post-operative weight-bearing instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Boylan, MBA, Study Director — Zimmer Biomet
Locations (3):
- United States (3):
  - Eskenazi Health, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Inova Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | THP Hip Fracture Plating System
Started | 1
Completed | 0
Not Completed | 1
Not completed — Early Study Termination | 1

BASELINE CHARACTERISTICS:
Arm/Group | THP Hip Fracture Plating System
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 83 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Revision
Description: Revision rate due to device related complication(s) or non-union of the femur.
Time Frame: 6 weeks
Population: At the time of early study termination, 1 subject enrolled into the study; however, the only study completed follow-up visit was the 1-6 week visit.
Measure: Count of Participants; unit: Participants
Arm/Group | THP Hip Fracture Plating System
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Number of Participants With Radiographic Fracture Healing of the Femur (RUSH)
Description: Radiographic fracture healing as seen on x-ray and defined using Radiographic Union Score for Hips (RUSH) scoring system. The RUSH quantifies four measures of healing: cortical bridging, cortical fracture disappearance, trabecular consolidation, and trabecular fracture disappearance. Cortical healing is assessed in four anatomic femoral neck regions (anterior, posterior, medial, lateral) and trabecular healing is measured with two assessments (fracture line disappearance and consolidation of matrix). Each of the 10 assessed dimensions of radiographic femoral neck healing are scored 1 to 3, leading to a minimum score of 10 (no signs of healing) and a maximum score of 30 (perfect healing).
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | THP Hip Fracture Plating System
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Average FIX-IT Score (Clinical Fracture Healing of the Femur)
Description: The Function IndeX for Trauma (FIX-IT) score is an assessment tool for patients with lower extremity fractures, incorporating pain and the ability to weight-bear. The score utilizes two questions to assess the ability to bear weight and two questions to assess pain at the fracture site. The maximum subtotal for each set of questions is 6 points, yielding a maximum overall score of 12 points and a minimum score (lowest weight bearing and highest pain) of 0 points.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THP Hip Fracture Plating System
Number analyzed (Participants) | 1
score on a scale | 3 (0)

4. Secondary Outcome: Average EQ-5D-5L Score (Clinical Fracture Healing of the Femur)
Description: The EuroQol five dimensions questionnaire (EQ-5D-5L) is a five dimensional self-assessment that is comprised of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These five dimensions can be used to index a subject's health utility on a scale of 0 to 1, where 0 is death and 1 is perfect health. The scoring rule for EQ-5D permits scores less than 0, implying that some health states may be worse than death. The Health Status is scored on a VAS scale of 0 to 100, where 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine').
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THP Hip Fracture Plating System
Number analyzed (Participants) | 1
score on a scale
  6 weeks - Health Status | 75 (0)
  6 weeks - EQ-5D Score | .456 (0)

5. Secondary Outcome: Average VAS Pain Score
Description: VAS pain scale is a unidimensional measure of pain intensity. The pain VAS is a continuous scale comprised of a horizontal (HVAS) line, 10 centimeters (100 mm) in length. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THP Hip Fracture Plating System
Number analyzed (Participants) | 1
score on a scale | 16 (0)

ADVERSE EVENTS:
Time Frame: Per the protocol, ISO definitions were followed for adverse event data collection. All adverse events were captured for subjects enrolled through 12 months follow-up or study completion (including lost to follow-up), whichever came first. Only (1) subject was enrolled in this study and they completed their 1-6 week follow-up visit, thus adverse event data only exists through the 1-6 week follow-up visit.
Description: ISO definition is not materially different from clinicaltrials.gov definitions.
Arm/Group | THP Hip Fracture Plating System
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THP Hip Fracture Plating System (N=1)
Dysphagia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT03870477/Prot_SAP_000.pdf